CLINICAL TRIAL: NCT06707090
Title: A Phase 3 Randomized, Parallel Group, Double-Blind Study to Evaluate the Efficacy, Tolerability, and Safety of TR987® 0.1% Gel Versus Standard of Care in the Treatment of Chronic Venous Insufficiency Leg Ulcers (VLU)
Brief Title: Tissue Repair Gel in Venous Leg Ulcers (US)
Acronym: TRIVIA
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: TR Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BG002
Record Dates: First submitted 2024-11-24; First posted 2024-11-27 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-09

CONDITIONS: Venous Leg Ulcer; Venous Ulcer; Venous Stasis Ulcer; Venous Stasis; Wound Heal; Wounds; Venous Insufficiency of Leg; Non-healing Wound
Keywords: Tissue Repair; Glucoprime; TR Therapeutics; Debridement; VLU
MeSH Terms: conditions — Varicose Ulcer; Wounds and Injuries | interventions — Gels; Standard of Care

STUDY DESIGN:
Intervention Model Description: This is an outpatient, randomized, parallel- group, double-blind, multicenter, 16-week study with 2 treatment arms: TR987 0.1% gel + Standard of Care and Standard of Care alone in participants who have a non-healing Venous Leg Ulcer (VLU)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants will be randomized to either TR987 1% gel + Standard of Care and Standard of Care alone. Sponsor, participant, and Investigator/Outcomes Assessor will be masked throughout the treatment period.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TR987 0.1% gel + Standard of Care (Experimental): Participants will receive up to 16 weeks of TR987 0.1% gel topically + Standard of Care (wound cleansing/dressings and compression bandaging). Treatment will be twice weekly for the first four weeks then weekly for the remaining 12 weeks.
  Interventions: Drug: TR987 0.1% gel + Standard of Care
- Standard of Care (Other)
  Interventions: Other: Standard of care

INTERVENTIONS:
Drug: TR987 0.1% gel + Standard of Care — 6mg topical gel for application plus Standard of Care (wound cleansing/dressings and compression bandaging)
  Arms: TR987 0.1% gel + Standard of Care
Other: Standard of care — Standard of Care (wound cleansing/dressings and compression bandaging)
  Arms: Standard of Care

SUMMARY:
The goal of this clinical trial is to learn if TR987 0.1% gel + Standard of Care works better than Standard of Care alone to treat Venous Leg Ulcers (VLUs). It will also provide additional information about the safety of drug TR987 0.1% gel.

DETAILED DESCRIPTION:
This is an outpatient, randomized, parallel- group, double-blind, multicenter, 16-week study with 2 treatment arms: TR987 0.1% gel + Standard of Care and Standard of Care alone in participants who have a non-healing Venous Leg Ulcer (VLU).

The primary objective is to assess the proportion of participants with Complete Closure of the target ulcer at or before the Week-16 end of treatment (EOT) visit.

Secondary endpoints include: • Proportion of participants with Complete Closure of the target ulcer at or before the Week 16 visit AND for whom the ulcer remains closed at the 3-Month Follow-Up visit after such closure (a composite endpoint). • Change from baseline in participant's perception of pain level at 12 weeks. • Percent change from baseline in the target ulcer area at 12 and 16 weeks. In the event of Complete Closure before these time points, the target ulcer area will be deemed to be zero at those time points for purposes of calculation of this endpoint. • Proportion of participants with Complete Closure of the target ulcer at or before the Week 12 treatment visit. • Proportion of participants with any significant reduction in pain at or before 12 weeks. There are also some supplementary and safety endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years and older
* Venous insufficiency has been clinically diagnosed clinically and medically confirmed.
* Females who are neither pregnant nor breastfeeding and if of child-bearing potential are on an acceptable method of birth control.
* The Venous Ulcer should be between 2 cm2 and 12 cm2 at randomization.
* Target ulcer age must be ≥ 4 weeks at Screening.
* Participants must have adequate arterial flow as confirmed by ABI/TBI, TB, SPP, TCPo2, or Duplex Doppler.
* Body mass index (BMI) ≤ 50 kg/m2.
* HbA1C ≤12%.

Exclusion Criteria:

* Target ulcer has been treated with prohibited medications or therapies.
* History of radiation at the target ulcer site.
* Target ulcer decreases in area by 30% or more during screening period.
* History of osteomyelitis at the target ulcer within 6 months of screening.
* Participants considered nutritionally deficient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 312 (Estimated)
Dates: Start 2025-01-28 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with Complete Closure of the target ulcer at or before the Week-16 end of treatment (EOT) visit. | 16 weeks
  Patient count

SECONDARY OUTCOMES:
Proportion of participants with Complete Closure of the target ulcer at or before the Week 16 visit AND for whom the ulcer remains closed at the 3-Month Follow-Up visit after such closure (a composite endpoint) | 16 weeks
  Patient count
Change from baseline in participant's perception of pain level at 12 weeks. | 12 weeks
  Pain to be measured on a 10 point numeric rating scale
Percent change from baseline in the target ulcer area at 12 and 16 weeks. In the event of Complete Closure before these time points, the target ulcer area will be deemed to be zero at those time points for purposes of calculation of this endpoint. | 12 and 16 weeks
  Measure the are of the wound in cm2 at baseline and at 12 and 16 weeks and calculate the percentage change
Proportion of participants with Complete Closure of the target ulcer at or before the Week 12 treatment visit. | 12 weeks
  Count the number of patients with complete closure and divide by the total number of patients
Proportion of participants with any significant reduction in pain at or before 12 weeks. | 12 weeks
  Count the number of patients with any significant reduction in pain and divide by the total number of patients
Proportion of target ulcers which reach greater than 70% closure at 12 weeks and 16 weeks | 12 and 16 weeks
  Measured by MolecuLight® versus baseline area at TV1 after therapeutic debridement (Complete Closure at a time point before 12 or 16 weeks shall be deemed to be >70% closed at 12 or 16-weeks, respectively, for purposes of this analysis)
Proportion of target ulcers which reach greater than 90% closure at 12 weeks and 16 weeks | 12 and 16 weeks
  Measured by MolecuLight® versus baseline area at TV1 after therapeutic debridement (Complete Closure at a time point before 12 or 16 weeks shall be deemed to be >70% closed at 12 or 16-weeks, respectively, for purposes of this analysis)
Proportion of target ulcers which reach greater than 95% closure at 12 weeks and 16 weeks | 12 and 16 weeks
  Measured by MolecuLight® versus baseline area at TV1 after therapeutic debridement (Complete Closure at a time point before 12 or 16 weeks shall be deemed to be >70% closed at 12 or 16-weeks, respectively, for purposes of this analysis)

CONTACTS AND LOCATIONS:
Locations (33):
- United States (33):
  - Clincial Research Site 21, Tucson, Arizona
  - Clincial Research Site 43C, Castro Valley, California
  - Clincial Research Site 14, Fresno, California
  - Clincial Research Site 11, Los Angeles, California
  - Clincial Research Site 43A, San Francisco, California
  - Clincial Research Site 43B, San Francisco, California
  - Clincial Research Site 54, Vista, California
  - Clincial Research Site 47, Deerfield Beach, Florida
  - Clincial Research Site 38, Hollywood, Florida
  - Clincial Research Site 40, Jacksonville, Florida
  - Clincial Research Site 19, Miami, Florida
  - Clincial Research Site 26, Miami, Florida
  - Clincial Research Site 13, Pembrook Pines, Florida
  - Clincial Research Site 51, Tamarac, Florida
  - Clincial Research Site 22, Chicago, Illinois
  - Clincial Research Site 34, Chicago, Illinois
  - Clincial Research Site 10, O'Fallon, Illinois
  - Clincial Research Site 49, Springfield, Illinois
  - Clincial Research Site 04, Bossier City, Louisiana
  - Clincial Research Site 01, Lafayette, Louisiana
  - Clincial Research Site 07, D'Iberville, Mississippi
  - Clincial Research Site 02, McComb, Mississippi
  - Clincial Research Site 30, New York, New York
  - Clincial Research Site 37, Syosset, New York
  - Clincial Research Site 55, Winston-Salem, North Carolina
  - Clincial Research Site 45, Grove City, Ohio
  - Clincial Research Site 23, Mentor, Ohio
  - Clincial Research Site 28, Tulsa, Oklahoma
  - Clincial Research Site 36, Philadelphia, Pennsylvania
  - Clincial Research Site 24, Fort Worth, Texas
  - Clincial Research Site 32, Houston, Texas
  - Clincial Research Site 46, San Antonio, Texas
  - Clincial Research Site 18, Suffolk, Virginia

IPD SHARING:
Plan to Share IPD: No
If the clinical data will be published, the relevant information may be made available.

REFERENCES:
- See also: Related Info — https://www.triviastudy.com